CLINICAL TRIAL: NCT03406585
Title: A Double-blinded, Randomized, Placebo-controlled Trial With Wharton's Jelly Derived Allogeneic Mesenchymal Stromal Cells (WJMSCs) for Preserving Endogenous Insulin Production in Adult Patients Diagnosed for Type 1 Diabetes
Brief Title: Wharton´s Jelly Derived Mesenchymal Stromal Cell Treatment of Adult Patients Diagnosed With Type I Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NextCell Pharma Ab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProTrans-T1D; 2017-002766-50 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2018-01-23 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic transplantation with WJMSCs (Experimental): Single infusion of 200 million cells per patient.
  Interventions: Drug: ProTrans: Allogeneic transplantation with WJMSCs
- Sham transplantation (placebo) (Placebo Comparator): Single infusion with albumin and dmso in sodium chloride (identical concentrations as active treatment)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ProTrans: Allogeneic transplantation with WJMSCs — The drug is a cell suspension with allogeneic mesenchymal stromal cells derived from umbilical cord tissue.
  Other Names: Protrans
  Arms: Allogeneic transplantation with WJMSCs
Drug: Placebos — Placebo treatment
  Other Names: Placebo
  Arms: Sham transplantation (placebo)

SUMMARY:
To investigate the safety and tolerance after allogeneic infusion of WJMSCs intravenously in adult patients diagnosed with type 1 diabetes.

DETAILED DESCRIPTION:
This is a combined phase I and phase II study, where the first part is an open, dose escalating study consisting of 9 male patients, 18-40 years of age. The second part is a randomized, double-blinded, placebo-controlled, phase I/II study in parallel design comparing allogeneic WJMSC treatment to placebo in adult patients diagnosed with type 1 diabetes. Besides safety, preservation of endogenous insulin production (measured as C-peptide concentrations) together with metabolic control, diabetes treatment satisfaction and immunological profile will be assessed.

A total number of 24 patients will be enrolled in the study and followed for one year after WJMSC/placebo treatment. Patients 18-40 years of age, both male and female, diagnosed for type 1 diabetes will be eligible. Providing informed consent and fulfillment of inclusion criteria and no exclusion criteria, they will within two years of diagnosis be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation of the study, given before undergoing any study-specific procedures
2. Clinical history compatible with type 1 diabetes diagnosed less than 2 years before enrolment
3. In the first part of the study patients 1-9 only male patients between 18-40 years of age will be included. In the second part of the study, patients 10-24, both male and female patients 18 to 40 years of age (inclusive at both ends) will be included.
4. Mentally stable and, in the opinion of the investigator, able to comply with the procedures of the study protocol
5. Fasting plasma C-peptide concentration >0.12 nmol/L.
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, if they are using effective methods of contraception during the study. Acceptable birth control methods are those with a failure rate of less than 1% per year when used consistently and correctly. Such methods include (in "Recommendations related to contraception and pregnancy testing in clinical trials", supplied from www.hma.eu/):

   1. Combined (estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation.

      * oral
      * intravaginal
      * transdermal
   2. progestogen-only hormonal contracption associated with inhibition of ovulation

      * oral
      * injectable
      * implantable
   3. intrauterine device (IUD)
   4. intrauterine hormone-releasing system (IUS)
   5. bilateral tubal occlusion
   6. total abstinence or vasectomized partner.

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients with body mass index (BMI) > 30, or weight >100 kg
3. Patients with weight <50 kg
4. Patients with unstable cardiovascular status incl. NYHA class III/IV or symptoms of angina pectoris.
5. Patients with uncontrolled hypertension (≥160/105 mmHg).
6. Patients with active on-going infections.
7. Patients with latent or previous as well as on-going therapy against tuberculosis, or exposed to tuberculosis or has travelled in areas with high risk of tuberculosis or mycosis within the last 3 months.
8. Patients with serological evidence of infection with HIV, Treponema pallidum, hepatitis B antigen (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.
9. Patients with any immune suppressive treatment
10. Patients with known demyelinating disease or with symptoms or physical examination findings consistent with possible demyelinating disease-
11. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
12. Patients with known, or previous, malignancy.
13. Taking oral anti-diabetic therapies or any other concomitant medication which may interfere with glucose regulation other than insulin.
14. Patients with GFR <80 ml/min/1.73 m2 body surface.
15. Patients with proliferative retinopathy.
16. Patient with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo treatment with MSC.
17. Known hypersensitivity against any excipients, i.e. dimethyl sulfoxide (DMSO).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Safety; measured through set safety parameters | throughout the study untill day 372
  measured through the registration of adverse events and other safety parameters such as hypoglycemia, allergic reactions, ophthalmologic examination, ECG, vital signs and laboratory assessments.
Efficacy; comparison of the intervention versus placebo at day 372 versus start of treatment | Day 372
  Delta-change of C-peptide Area Under the Curve (AUC) (0-120 min) for Mixed Meal Tolerance Test (MMTT) at day 372 following WJMSC/Placebo infusion when compared to test performed before start of treatment.

SECONDARY OUTCOMES:
Number of patients insulin independent (ADA criteria) at days 187 and 372 | Days 187 and 372 following WJMSC/Placebo infusion
  Insulin doses and measured plasma glucose values are written down in the subject's diary every day by the subject. Amount of insulin, recorded plasma glucose values, time and date will be included
Number of patients with daily insulin needs <0.25U/kg at days 187 and 372 | Days 187 and 372 following WJMSC/Placebo infusion
  Insulin doses and measured plasma glucose values are written down in the subject's diary every day by the subject. Amount of insulin, recorded plasma glucose values, time and date will be included
Insulin requirement/kg BW at days 187 and 372 | Days 187 and 372 following WJMSC/Placebo infusion
  Insulin doses and measured plasma glucose values are written down in the subject's diary every day by the subject. Amount of insulin, recorded plasma glucose values, time and date will be included
HbA1c at days 187 and 372. | Days 187 and 372 following WJMSC/Placebo infusion
  Measurements of HbA1c will be performed to assess metabolic control during study.
Glucose variability at day 372 | Day 372 following WJMSC/Placebo infusion
  Measurements of HbA1c will be performed to assess metabolic control during study.
Delta change of levels of fasting C-peptide at day 372 | Day 372 following WJMSC/Placebo infusion
  Measured at day 372 compared to before start of treatment
Numbers of patients with peak C-peptide >0.20 nmol/l, in response to the MMTT, at day 372 | Day 372 following WJMSC/Placebo infusion
  Measured at day 372 compared to before start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — NextCell Pharma
Locations (1):
- Karolinska Trial Alliance, Fas 1 enheten, Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlsson PO, Espes D, Sisay S, Davies LC, Smith CIE, Svahn MG. Umbilical cord-derived mesenchymal stromal cells preserve endogenous insulin production in type 1 diabetes: a Phase I/II randomised double-blind placebo-controlled trial. Diabetologia. 2023 Aug;66(8):1431-1441. doi: 10.1007/s00125-023-05934-3. Epub 2023 May 24. PMID 37221247